CLINICAL TRIAL: NCT01300637
Title: Prevalence of Metabolic Syndrome and Effects of Adjunctive Metformin on Metabolic Profiles in Clozapine-treated Schizophrenic Patients
Brief Title: Effects of Adjunctive Metformin on Metabolic Profiles in Clozapine-treated Schizophrenic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chun-Hsin Chen, Taipei Medical University-WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 96064
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Obesity; Metabolic Syndrome; Schizophrenia
Keywords: schizophrenia; clozapine; metabolic dysregulation; metformin
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Schizophrenia | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin (Active Comparator): metformin intervention group
  Interventions: Drug: Metformin
- placebo (Placebo Comparator): placebo-controlled
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metformin — metformin 500 mg/pill; target dose 1500 mg/day for 24 weeks
  Other Names: Diaformin 500 mg/pill
  Arms: metformin
Drug: placebo — identical-appearing pill of placebo
  Other Names: Diaformin 500 mg/pill identical-appearing placebo
  Arms: placebo

SUMMARY:
Background: Several studies have suggested that clozapine has the greatest propensity of all available atypical antipsychotics to induce weight gain and metabolic dysregulation. So it is necessary to conduct some interventions to prevent or treat metabolic dysregulation induced by clozapine.

Metformin has been reported to achieve weight loss in several groups of patients characterized by insulin resistance. Several studies evaluated the effects of metformin on antipsychotics-induced weight gain and study period lasted from 8 to 16 weeks. Long-term metformin use had more robust effect on metabolic dysregulation and body weight in non-psychiatric field.

Goals: The study goals are two-fold. The first goal is to estimate the prevalence of metabolic dysregulation among clozapine-treated schizophrenic patients in Taiwan. The second goal is to assess the reversal effect of metformin on metabolic disturbance among clozapine-treated schizophrenic patients in a 24-week double-blind, placebo-control trial. The investigators will use metformin 1500 mg/d or placebo in the second phase trial.

Methods: This study will be divided into two phases. The first phase is to estimate the prevalence of metabolic disturbances among clozapine-treated patients. The second will be a randomized, double-blind, and placebo-controlled study of adjunctive metformin for non-DM clozapine-treated patients.

The clozapine dosage was maintained unchanged during the study period. The eligible patients will be randomly assigned to either metformin or identical placebo pills. Metformin will be titrated to 1500 mg/day in 4 weeks. Patients' blood pressure (BP), waist circumference, body weight, fasting plasma glucose (FPG), triglyceride (TG), high-density lipoprotein cholesterol (HDL), insulin, and leptin will be measured at 2, 4, 8, 16, and 24 weeks after the start of metformin.

In a 3-year period, the investigators estimate to recruit 150 clozapine-treated patients in the first phase and 75 fulfill the second phase criteria. The investigators estimate 60 patients complete the second phase intervention (staying in second phase at least 4 weeks).

From this study, the investigators would like to know the prevalence of metabolic dysregulation among clozapine-treated schizophrenic patients and to know the effect of metformin on metabolic profile among non-DM clozapine treated patients.

DETAILED DESCRIPTION:
Background: Several studies have suggested that clozapine has the greatest propensity of all available atypical antipsychotics to induce weight gain and metabolic dysregulation. So it is necessary to conduct some interventions to prevent or treat metabolic dysregulation induced by clozapine.

Metformin has been reported to achieve weight loss in several groups of patients characterized by insulin resistance. Several studies evaluated the effects of metformin on antipsychotics-induced weight gain and study period lasted from 8 to 16 weeks. Long-term metformin use had more robust effect on metabolic dysregulation and body weight in non-psychiatric field. In our recent study data showed that after 8 weeks treatment with metformin 1500 mg/day in 24 olanzapine-treated patients, the body weight, fasting levels of glucose, triglyceride, and insulin significantly decreased. Insulin secretion and insulin resistance also decreased significantly. Half of subjects with metabolic syndrome obtained improvement after metformin trial.

Goals: The study goals are two-fold. The first goal is to estimate the prevalence of metabolic dysregulation among clozapine-treated schizophrenic patients in Taiwan. The second goal is to assess the reversal effect of metformin on metabolic disturbance among clozapine-treated schizophrenic patients in a 24-week double-blind, placebo-control trial. We will use metformin 1500 mg/d or placebo in the second phase trial.

Methods: This study will be divided into two phases. The first phase is to estimate the prevalence of metabolic disturbances among clozapine-treated patients. The second will be a randomized, double-blind, and placebo-controlled study of adjunctive metformin for non-DM clozapine-treated patients.

Patients are recruited in the first phase if they meet the following criteria (1) fulfilled DSM-IV criteria of schizophrenia or schizoaffective disorder; (2) 18-65 year of age (3) receiving clozapine for at least 6 months. We will check patients' blood pressure (BP), waist circumference, body weight, fasting plasma glucose (FPG), triglyceride (TG), high-density lipoprotein cholesterol (HDL), insulin, and leptin will be measured. In this study, we use the modified ATP III criteria for Asians to evaluate subjects for a diagnosis of metabolic syndrome.

The inclusion criteria of second phase intervention will be first-phase participants who are (1) overweight and obese (BMI ≧ 24) or (2) one or more metabolic dysregulation, such as abdominal obesity (waist circumference > 90 cm, in men and > 80 cm, in women; fasting hypertriglyceridemia, (≥ 150 mg/dL); low fasting HDL levels (< 40 mg/dL in men and < 50 mg/dL in women); high blood pressure (≥ 130/ ≥ 85 mm Hg or current treatment with antihypertensive medication). The exclusion criteria are the following: (1) current use of hypoglycemic or hypolipidemic agents (2) FPG levels ≥ 126 mg/dL; (3) women who are pregnant; (4) known allergy or contraindicated to metformin (including Creatine>1.4 ng/dl; abnormal liver function test; chronic cardiopulmonary insufficiency).

The clozapine dosage was maintained unchanged during the study period. The eligible patients will be randomly assigned to either metformin or identical placebo pills. Metformin will be titrated to 1500 mg/day in 4 weeks. Patients' blood pressure (BP), waist circumference, body weight, fasting plasma glucose (FPG), triglyceride (TG), high-density lipoprotein cholesterol (HDL), insulin, and leptin will be measured at 2, 4, 8, 16, and 24 weeks after the start of metformin.

In a 3-year period, we estimate to recruit 150 clozapine-treated patients in the first phase and 75 fulfill the second phase criteria. We estimate 60 patients complete the second phase intervention (staying in second phase at least 4 weeks).

From this study, we would like to know the prevalence of metabolic dysregulation among clozapine-treated schizophrenic patients and to know the effect of metformin on metabolic profile among non-DM clozapine treated patients.

Key words: schizophrenia, clozapine, metabolic dysregulation, metformin

ELIGIBILITY:
Inclusion Criteria:

phase 1

* fulfilled DSM-IV criteria of schizophrenia or schizoaffective disorder
* 18-65 year of age
* receiving clozapine for at least 6 months.

phase 2 are those in phase 1 and met the following

* overweight and obese (BMI ≧ 24)
* one or more metabolic dysregulation, such as abdominal obesity (waist circumference > 90 cm, in men and > 80 cm, in women
* fasting hypertriglyceridemia, (≥ 150 mg/dL)
* low fasting HDL levels (< 40 mg/dL in men and < 50 mg/dL in women)
* high blood pressure (≥ 130/ ≥ 85 mm Hg or current treatment with antihypertensive medication).

The exclusion criteria are the following:

* current use of hypoglycemic or hypolipidemic agents
* FPG levels ≥ 126 mg/dL
* women who are pregnant
* known allergy or contraindicated to metformin (including Creatine>1.4 ng/dl abnormal liver function test; chronic cardiopulmonary insufficiency).

Exclusion Criteria:

phase 2

* current use of hypoglycemic or hypolipidemic agents
* FPG levels ≥ 126 mg/dL
* women who are pregnant
* known allergy or contraindicated to metformin (including Creatine>1.4 ng/dl abnormal liver function test
* chronic cardiopulmonary insufficiency).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-04 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
body weight change | 24 weeks
  We measure body weight before and after intervention, at week 2, 4, 8, 16, 24

SECONDARY OUTCOMES:
metabolic features | 24 weeks
  Our secondary outcomes included waist circumference, blood pressure, triglyceride, HDL-C, fasting glucose and insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hsin Chen, MD, Principal Investigator — Taipei Medical University-WanFang Hospital, Taipei, Taiwan
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen CH, Huang MC, Kao CF, Lin SK, Kuo PH, Chiu CC, Lu ML. Effects of adjunctive metformin on metabolic traits in nondiabetic clozapine-treated patients with schizophrenia and the effect of metformin discontinuation on body weight: a 24-week, randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2013 May;74(5):e424-30. doi: 10.4088/JCP.12m08186. PMID 23759461